CLINICAL TRIAL: NCT04037995
Title: Real World Study of End-stage Liver Disease in China
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Chief of dpartment of infectious disease, Huashan Hospital
Other Study IDs: KY2019-RWS(LD)
Record Dates: First submitted 2019-07-14; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: End Stage Liver DIsease; Complication
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervation — No intervation

SUMMARY:
The aims of this study are exploring the current situation of end-stage liver disease in China, and the optimization of diagnosis and treatment. Liver cirrhosis often accompanied by a series of complications. Therefore, it is necessary to standardize the diagnosis and treatment of liver cirrhosis and its complications. End-stage liver disease mainly refers to the late stage of liver disease caused by various chronic liver damage. Its main feature is that liver function can not meet the physiological needs of human body. This study is a single-center, prospective and observational real-world study aimed at investigating and analyzing the current diagnosis and treatment of liver cirrhosis and end-stage liver disease in China.

DETAILED DESCRIPTION:
The aims of this study are exploring the current situation of end-stage liver disease in China, and the optimization of diagnosis and treatment. Liver cirrhosis includes cirrhosis caused by hepatitis, alcoholic cirrhosis, non-alcoholic cirrhosis and schistosomiasis cirrhosis. Liver cirrhosis often accompanied by a series of complications, including portal hypertension and gastrointestinal bleeding, ascites and related infections, hepatorenal syndrome, hepatic encephalopathy, portal vein thrombosis, etc. Therefore, it is necessary to standardize the diagnosis and treatment of liver cirrhosis and its complications, but there are still disputes about most of the complications in various editions of the guidelines. In order to formulate the best empirical treatment plan, it is indispensable to master the epidemiological situation of cirrhosis in different places. However, there is a lack of support from large clinical data from China. End-stage liver disease mainly refers to the late stage of liver disease caused by various chronic liver damage. Its main feature is that liver function can not meet the physiological needs of human body. It covers the final stages of various chronic liver diseases, mainly manifested as severe impairment and decompensation of liver function, including chronic and acute liver failure, acute decompensation of cirrhosis, chronic liver failure and hepatocellular carcinoma. The concept of end-stage liver disease was first put forward in the 1980s and has not been strictly defined yet. However, due to the complications of end-stage liver disease, such as infection related to liver failure and portal hypertension, septic shock, hepatic encephalopathy, and serious decline in quality of life, and the one-year survival rate of most patients is less than 90%, it is necessary to put forward this concept. Therefore, there is still a need for large sample data to define end-stage liver disease and formulate evidence-based treatment plans.

The aim of this study is to explore the efficacy, safety and economic benefits of different treatment options for patients with cirrhosis and complications and end-stage liver disease in the real world of China. To investigate the epidemiological rates of cirrhosis and end-stage liver disease, and to provide evidence-based medical evidence for the treatment and follow-up of cirrhosis and end-stage liver disease in China in the future.

This study is a single-center, prospective and observational real-world study aimed at investigating and analyzing the current diagnosis and treatment of end-stage liver disease in China, exploring the situation of end-stage liver disease in China, exploring the treatment options for patients with end-stage liver disease that can effectively improve their prognosis, and seeking high-quality evidence-based medical treatment for cirrhosis and reducing the mortality of end-stage liver disease.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent of patients.
2. Diagnosis of any of the following diseases: acute decompensation of cirrhosis, chronic and acute liver failure, chronic liver failure and hepatocellular carcinoma (stage III-IV)

Exclusion Criteria:

1. HIV antibody positive and AIDS patients
2. Serious psychiatric history, especially depression. Severe mental illness is defined as major depression or psychosis, suicide attempts, hospitalization due to mental illness or a period of disability due to mental illness.
3. Patients with serious diseases of heart, lung, kidney, brain, blood and other important organs.
4. Patients with other malignant tumors (excluding those cured).
5. Pregnant, lactating women or women of childbearing age who are ready to conceive.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population who were diagnosed of acute decompensation of cirrhosis, chronic and acute liver failure, chronic liver failure or hepatocellular carcinoma (stage III-IV)
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Patient died during follow-up | 3 years
  Death occurred during 3 year

SECONDARY OUTCOMES:
Major events occurred during follow-up | 3 years
  the major events including liver transplantation and the happening of serious complications

CONTACTS AND LOCATIONS:
Locations (1):
- HuaShan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] GBD 2016 Causes of Death Collaborators. Global, regional, and national age-sex specific mortality for 264 causes of death, 1980-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1151-1210. doi: 10.1016/S0140-6736(17)32152-9. PMID 28919116